CLINICAL TRIAL: NCT00351923
Title: Open, Multicenter, Randomised, Controlled Phase IIIb Study Evaluating the Immunogenicity and Safety of Subcutaneous Versus Alternative Administration Route of Combined MeMuRu-OKA Vaccine to Healthy Children Aged 11 to 21 Months.
Brief Title: Immunogenicity/Safety of Measles-Mumps-Rubella-Varicella Vaccine (MeMuRu-OKA): Using Two Different Administration Routes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106670
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox

INTERVENTIONS:
Biological: MeMuRu-OKA (study vaccine)

SUMMARY:
This study will compare the immunogenicity and safety of the MeMuRu-OKA vaccine administered subcutaneously or using an alternative administration route.

ELIGIBILITY:
Inclusion Criteria:

* Children must be healthy and have a birth weight > 2000 g to participate

Exclusion Criteria:

* confirmed or suspected tuberculosis, immunosuppressive (including HIV) conditions, neurological disorders, history of allergic disease or reaction, major congenital defects, chronical administration of salicylates, and fever (axillary temperature ³ 37.5°C at the time of vaccination) are excluding factors.
* Children from pregnant mothers who have a negative history of chickenpox are also excluded from the study.
* Children must have received one dose (but not more) of MMR and of varicella at least 6 weeks before entering the study. They must not receive or have received other non-registered drug or vaccine within 30 days prior to study start, or immunosuppressants for more than 14 days.
* Immunoglobulins or any blood products are prohibited during the 6 months before and during the study, as well as vaccine other than that foreseen by the protocol within 30 days before vaccination.
* Children must not have had measles, mumps, rubella or varicella/zoster, or have been exposed to those diseases within 30 days prior to study start.
* New-born infants (< 5 weeks of age), pregnant women without previous exposure to chickenpox, and immunodeficient persons cannot live in the same household as the vaccinated child

Ages: 11 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates after vaccination

SECONDARY OUTCOMES:
Antibody titres; safety: solicited local/ general, unsolicited AEs (42 days), SAEs (whole study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- Germany (18):
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate